CLINICAL TRIAL: NCT01759927
Title: Investigating the Effectiveness of Exercise Coaching on the Physical Activity Behavior of Physically Inactive Employees in a Company in Flanders: a Randomized Control Trial.
Brief Title: Investigating the Effectiveness of Exercise Coaching on the Physical Activity Behavior of Physically Inactive Employees.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Janssen Pharmaceutica (Industry)
Responsible Party: Principal Investigator, Jan Seghers, Principal Investigator, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S54788
Record Dates: First submitted 2012-12-30; First posted 2013-01-03 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Sedentary Lifestyle
Keywords: Physical activity counselor; Workplace intervention; Active and healthy lifestyle
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control condition (No Intervention): Physically inactive employees are measured on anthropometrics, fitness and psycho-social variables.
- Physical Activity Coaching (Experimental): Physically inactive employees receiving a 12-week behavioural support intervention grounded in self-determination theory.
  Interventions: Behavioral: physical activity coaching

INTERVENTIONS:
Behavioral: physical activity coaching — After measuring physical actity, physical fitness level, anthropometric and psychosocial variables a personalized 12 week physical activity program is made (=baseline). The intervention consisted of two face-to-face counselling sessions at the start of the intervention, short contacts by e-mail or telephone at weeks 3, 6 and 9, and two face-to-face counselling sessions at the end of the intervention. Employees exercise on their own. After 12 weeks and 6 months all measures are repeated.
  Arms: Physical Activity Coaching

SUMMARY:
The primary aim of this study is to investigate if and how a physical activity counselor can offer an added value in exercise promotion in physically inactive employees. We will explore if the physical activity counselor in the workplace setting can motivate sedentary employees to engage into systematic participation in sports and/or exercise by means of a short term coaching of 12 weeks. We aim to include 300 employees in the physical activity coaching process.

DETAILED DESCRIPTION:
Being physically active on a regular basis has many health benefits. Nevertheless, the majority of the Belgian population doesn't reach the recommended amount and intensity of physical activity to profit from these health benefits. A physical activity counselor can possibly play a crucial role for these physically inactive individuals. He/she can design an individualized exercise program to stimulate the person to become lifelong physical active. Research has shown that exercise promotion at work can result in a lower absenteeism, prevention of burn-out and a positive corporate identity.

ELIGIBILITY:
Inclusion Criteria:

* Employee of Janssen Pharmaceutics Belgium
* Physically inactive lifestyle (not reaching 150 minutes of moderate-to-vigorous physical activity a week)
* PAR-Q questionnaire all answers negative, if one or more answers are positive a permission of a physician is necessary

Exclusion Criteria:

* none

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2013-02; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in objective measure of degree of physical activity | baseline, 12 weeks, 6 months
  Sensewear: accelerometer worn on the upper arm during 7 consecutive days measuring the physical activity pattern during this period

SECONDARY OUTCOMES:
Change in health-related anthropometric measures | baseline, 12 weeks, 6 months
  Weight, Abdominal circumference, Bodycomposition (fat- and musclepercentage)

OTHER OUTCOMES:
Change in psycho-social variables | baseline, 12 weeks, 6 months
  Measuring general and work related well-being, motivation to be physically active and social identification with the physical activity group

CONTACTS AND LOCATIONS:
Overall Officials: Jan Seghers, Dr, Principal Investigator — Faculty of Kinesiology and Rehabilitation Sciences
Locations (1):
- Katholieke Universiteit Leuven - Faculty of Kinesiology and Rehabilitation Sciences, Leuven, Vlaams Brabant, Belgium

REFERENCES:
- [Derived] Arrogi A, Schotte A, Bogaerts A, Boen F, Seghers J. Increasing Employees' Health by Workplace Physical Activity Counseling: The Mediating Role of Step-Based Physical Activity Behavior Change. J Phys Act Health. 2019 Mar 1;16(3):205-213. doi: 10.1123/jpah.2018-0148. Epub 2019 Feb 15. PMID 30764729
- [Derived] Arrogi A, Schotte A, Bogaerts A, Boen F, Seghers J. Short- and long-term effectiveness of a three-month individualized need-supportive physical activity counseling intervention at the workplace. BMC Public Health. 2017 Jan 9;17(1):52. doi: 10.1186/s12889-016-3965-1. PMID 28069016